CLINICAL TRIAL: NCT00256516
Title: Low Carbohydrate Portfolio or "Eco-Atkins" Diet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 05-025
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Hypercholesterolemia; Cardiovascular Diseases
Keywords: Diet Therapy
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases

ARMS (2):
- Eco-Atkins diet (Experimental)
  Interventions: Other: Eco-Atkins diet (high vegetable protein and vegetable fat)
- NCEP diet (Active Comparator)
  Interventions: Other: NCEP diet

INTERVENTIONS:
Other: Eco-Atkins diet (high vegetable protein and vegetable fat)
  Arms: Eco-Atkins diet
Other: NCEP diet
  Arms: NCEP diet

SUMMARY:
Exchange of the butter, eggs, cheese and meat in the Atkins diet for soy protein foods, other vegetable proteins including gluten and vegetable fats, nuts, avocado, olive and canola oil will result in dramatic rather than modest reductions in blood lipids with weight loss. In effect this will represent an exchange of saturated fat and animal protein for healthy monounsaturated and polyunsaturated fats and vegetable proteins with significant effects on blood lipids while still encouraging weight loss.

DETAILED DESCRIPTION:
Subjects: Thirty overweight hyperlipidemic subjects who wish to lose weight.

Design:

* Protocol (Metabolic Study): will be randomized to either the Eco-Atkins diet (15 subjects) or NCEP diet (15 subjects). The diets will be provided for the one month period with the aim of inducing the same weight loss (5 kg) as seen in the first month of the published reports on the Atkins diet. The diets will provide about 60% of estimated energy requirements. Subjects will be provided with their diets at weekly intervals by courier and intakes adapted to ensure that they achieve their target weight loss goal. Fasting weight will be taken at weekly intervals together with blood pressure and blood for lipids, glucose and insulin assessment.
* Protocol (Ad Libitum Study): After completing the metabolic phase of the study, the thirty subjects will be asked to continue with the diet to which they were randomized for a further 6-month period. During this ad libitum trial, study foods will not be provided. This longer less tightly controlled study will establish the value of this diet in "real life" situations. This will be required to support our shorter term, well-controlled more detailed metabolic study. Fasting weight will be taken at monthly intervals together with blood pressure and blood for lipids, glucose and insulin assessment.

Study Details: Participants will come after a 12h overnight fast to the Risk Factor Modification Centre at St. Michael's Hospital or the Department of Nutritional Sciences, University of Toronto immediately prior to commencement of each treatment phase and at weekly intervals during the metabolic study and monthly during the ad libitum study. Prior to the start of the study, participants will be instructed on details of the study diet protocol. They will also be asked to maintain a constant level of physical activity throughout the course of the study. At all visits, body weight (in kg) will be obtained in indoor clothing, without shoes, and blood pressure will be taken twice in the dominant arm after participants have been seated for at least 20 minutes. Height (in cm) will be recorded at the first visit. Body composition measurements will be measured using bioelectric impedance at baseline and week 4 of the metabolic phase, and months 3 and 6 of the ad libitum phase. Throughout the study period, participants will maintain the diet prescribed on their initial visit. At each visit, participants will provide a fasting blood sample and seven-day food records will be collected. During the last week of the metabolic and ad libitum study, 24h fecal and urine collections will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women between the age of 21 and 70
* Body mass index > 27 kg/m2 and whose body weight has remained constant over the last 6 months preceding the onset of the study.
* Fasting plasma LDL cholesterol concentration > 3.4 mmol/L at diagnosis.
* Treated by diet.
* Alcohol intake < 14 drinks per week.
* Fasting plasma triglyceride concentration > 0.5 mmol/L and < 5.0 mmol/L.
* Living within a 40 km radius of St. Michael's Hospital or the University of Toronto.

Exclusion Criteria:

* Premenopausal women due to the fluctuation of blood lipids during the menstrual cycle.
* Taking lipid lowering medications. (However, with their physician's approval those who wish to join but are already taking cholesterol-lowering medications may join the study providing the medications are stopped for at least two weeks before starting the study and throughout the study.)
* Evidence of major cardiovascular event (stroke or myocardial infarction) within the past 6 months.
* Positive molecular diagnosis of familial hypercholesterolemia.
* Secondary causes of hypercholesterolemia (hypothyroidism, renal or liver disease).
* Diabetes
* Uncontrolled high blood pressure (> 140/90mmHg).
* Major disability or disorder such as liver disease, renal failure or cancer or with major surgery < 6 months prior to randomization.
* LDL-C levels below 3.0 mmol/L on a Step 2 diet prior to randomization.
* Postmenopausal women on hormone replacement therapy
* Smokers
* Patients with food allergies.
* Patients with a history of any form of cancer or are considered at high risk for cancer. However, if such patients wish to join the study, we, the researchers, would like them to obtain the approval of their oncologist or responsible physician prior to enrollment in the study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Study Completion 2006-12

PRIMARY OUTCOMES:
total and low-density lipoprotein (LDL) cholesterol
LDL:HDL cholesterol ratio
weight reduction

SECONDARY OUTCOMES:
blood pressure
high-density lipoprotein (HDL) cholesterol
HDL2 and HDL3, triglyceride, apolipoprotein A1 and B, Lp(a) and LDL particle size
glucose, insulin and measurements of oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, PhD, DSc, Principal Investigator — University of Toronto and St. Michael's Hospital
Locations (1):
- Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Jenkins DJ, Wong JM, Kendall CW, Esfahani A, Ng VW, Leong TC, Faulkner DA, Vidgen E, Greaves KA, Paul G, Singer W. The effect of a plant-based low-carbohydrate ("Eco-Atkins") diet on body weight and blood lipid concentrations in hyperlipidemic subjects. Arch Intern Med. 2009 Jun 8;169(11):1046-54. doi: 10.1001/archinternmed.2009.115. PMID 19506174
- [Derived] Jenkins DJ, Wong JM, Kendall CW, Esfahani A, Ng VW, Leong TC, Faulkner DA, Vidgen E, Paul G, Mukherjea R, Krul ES, Singer W. Effect of a 6-month vegan low-carbohydrate ('Eco-Atkins') diet on cardiovascular risk factors and body weight in hyperlipidaemic adults: a randomised controlled trial. BMJ Open. 2014 Feb 5;4(2):e003505. doi: 10.1136/bmjopen-2013-003505. PMID 24500611
- [Derived] Wong JM, Kendall CW, Marchie A, Liu Z, Vidgen E, Holmes C, Jackson CJ, Josse RG, Pencharz PB, Rao AV, Vuksan V, Singer W, Jenkins DJ. Equol status and blood lipid profile in hyperlipidemia after consumption of diets containing soy foods. Am J Clin Nutr. 2012 Mar;95(3):564-71. doi: 10.3945/ajcn.111.017418. Epub 2012 Feb 1. PMID 22301925